CLINICAL TRIAL: NCT00691691
Title: A Phase II Study of Fractionated Stereotactic Body Radiation Therapy (SBRT) in the Treatment of Liver Tumors
Brief Title: Stereotactic Body Radiation Therapy (SBRT) in the Treatment of Liver Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alberta Health services (Other)
Responsible Party: Dr. Robert Nordal, Tom Baker Cancer Centre
Organization: AHS Cancer Control Alberta (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18740; 18740
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2011-08

CONDITIONS: Liver Tumors
Keywords: Liver malignancy; Stereotactic Body Radiation Therapy; Efficacy of SBRT in liver tumors; Hepatic toxicity with SBRT
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Eligible patient will be treated with 48 Gy in 4 fractions encompassing the entire target lesion in 2 weeks with a minimum of 48 hours between each dose.
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — Radiation Dose: 48 Gy in 4 fractions in 2 weeks. A minimum of 48 hours should separate each treatment (e.g. every Tuesday and Friday). The dose is prescribed to the marginal isodose (80-90%) that encompasses the entire target lesion (GTV). Treatment will be delivered using a linear accelerator. For verification of the accuracy of these external skin fiducial markers, 10 patients will also have implanted internal gold coil markers. The implantable gold coil markers will be implanted into the liver in the proximity of the target lesions via a percutaneous transhepatic route under fluoroscopy guidance.

SUMMARY:
Patients with primary hepato-biliary malignancies or liver metastases from gastrointestinal cancer suffer substantial morbidity and mortality from their hepatic disease. Curative resection is feasible only for selected subgroups of patients. The majority of patients have unresectable and incurable disease. Aggressive arterial and systemic chemotherapy have been used in recent years with improved response and survival. However, a significant number of patients, at least one-third of patients with liver metastases from colorectal cancer and two-third or higher of unresectable hepatobiliary cancer, continue to die of liver failure from progressive disease in the liver. Percutaneous ethanol injections, chemoembolization, cryotherapy and thermal ablation using radiofrequency have been used to treat selected patients with smaller tumors (3-4 cm) in areas away from major blood vessels and the biliary tract. However, most unresectable liver cancers did not fit the criteria for these treatments. Therefore, other regional therapeutic option like external radiation therapy may be considered for local control in the liver or symptom palliation

ELIGIBILITY:
Inclusion Criteria:

* Histologically conformation of liver malignancy
* Solitary or multiple liver tumors amenable to SBRT
* No jaundice or liver dysfunction
* For metastases, the primary tumor site has been adequately treated.
* For primary hepatoma, no extra-hepatic disease
* Karnofsky > 70

Exclusion Criteria:

* no extra-hepatic disease
* Liver failure or inadequate liver function
* Ascites
* Previous radiation therapy to the liver
* lesions invading major blood vessels in the porta region
* Contraindication to receive radiation therapy in the liver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2007-11

PRIMARY OUTCOMES:
Response rate to SBRT | 3-6 Months

SECONDARY OUTCOMES:
Treatment Related Toxicity | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Nordal, M.D., Principal Investigator — Tom Baker Cancer Centre
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada